CLINICAL TRIAL: NCT03827031
Title: Implementation and Impact of Multidisciplinary Medication Review in Surgery Departments on Medication Management of Elderly Patients
Brief Title: Impact of Mulstidisciplinary Medication Assessment Review in Surgery Departments
Acronym: CHIROPMEV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NIMAO/2017-02/JMK-01
Record Dates: First submitted 2018-08-22; First posted 2019-02-01 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Chronic Disease
Keywords: Drug Safety; Clinical Pharmacy; General Practice; Surgery; Geriatrics; Medication Review
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (No Intervention)
- B1 interventional group (Experimental)
  Interventions: Other: Mutlidisciplinary medication Review (MMR)
- B2 interventional group (Experimental)
  Interventions: Other: Mutlidisciplinary medication Review (MMR); Other: Mutlidisciplinary medication Review (MMR) with community pharmacist follow-up

INTERVENTIONS:
Other: Mutlidisciplinary medication Review (MMR) — The clinical pharmacist performs medication reconciliation and pharmaceutical analysis. The physician performs a clinical examination and analysis of the medical record. Both participate in a collaborative interview. The hospital physician calls the community pharamcist to discuss proposed changes on the order and to establish a new prescription. At the end of the stay, the clinical pharmacist will conduct an exit interview with the patient. Three months after discharge, the patient's community pharmacist will be contacted to assess whether the changes proposed in the MMR were accepted
  Arms: B1 interventional group; B2 interventional group
Other: Mutlidisciplinary medication Review (MMR) with community pharmacist follow-up — Multidisciplinary medication review (MMR) The clinical pharmacist performs medication reconciliation and pharmaceutical analysis. The physician performs a clinical examination and analysis of the medical record. Both participate in a collaborative interview. The hospital physician calls the community physician to discuss proposed changes on the order and to establish a new prescription. At the end of the stay, the clinical pharmacist will conduct an exit interview with the patient.
  Community follow-up A summary of the follow-up report stating the therapeutic modifications (called below multidisciplinary correspondence documents) will be sent to the community pharmacist and physician. Within 2 months of discharge, the pharmacist performs a follow-up of medication changes accepted and not accepted by the community physician.
  Three months after discharge, the patient's community pharmacist will be contacted to assess whether the changes proposed in the MMR were accepted.
  Arms: B2 interventional group

SUMMARY:
The presence of a clinical pharmacist (for their pharmacological expertise) and a general practitioner (for their somatic expertise) in surgery departments would contribute to improve the management of medications in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* The patient (or their representative) has given his consent and signed the consent form.
* The patient is affiliated to a health insurance programme.
* The patient is at least 65 years old (≥) treated by at least (≥) five medications for at least (≥) 6 months
* The patient is available for a follow-up of 3 months.
* The patient is hospitalized in the surgery department.
* Patient with a Trivalle score greater than or equal to 2 (≥).
* Patient living in a nursing home or going back home after hospitalization.

Exclusion Criteria:

* The subject is participating in another category I interventional study.
* The subject is in an exclusion period determined by another study.
* The subject is under safeguard of justice.
* It is not possible to give the patient (or his/her trusted-person) informed information.
* Palliative care

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 297 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in iatrogenic drug risk in intervention groups versus control group | 3 months after hospitalization
  Proportion of patients transitioning from intermediate or high to low risk according to Trivalle score (a score between 0-10. A score 0-1 constitutes a low ADE risk (12%), score 2-5 represents an average risk (32%), and a score 6-10 represents a high risk (53%)

SECONDARY OUTCOMES:
Proportion of proposed medication modifications made by the clinical pharmacist accepted by the clinical doctor during the Multidisciplinary Medication Review in the experimental groups | Hospital discharge (maximum 30 days)
  Number of modifications accepted/number of modifications proposed
Number of potentially inappropriate medications per patient in each group | Hospital discharge (maximum 30 days)
Proportion of proposed medication modifications made by the collaborative team accepted and/or made permanent | 3 months after hospital discharge
  Number of modifications accepted/number of modifications proposed
Number of potentially inappropriate medications per patient in each group | 3 months after hospital discharge
Time required for Multidisciplinary Medication Review in the interventional groups (B1 and B2) | Hospital discharge (maximum 30 days)
  Hours
Time required for ransmitting multidisciplinary correspondence documents in B2 group | Hospital discharge (maximum 30 days)
  Hours
Number of multidisciplinary correspondence documents sent to the community acotors in B2 group | Hospital discharge (maximum 30 days)
Description of mode of diffusion of multidisciplinary correspondence documents in the B2 group | Hospital discharge (maximum 30 days)
  email, fax or letter
Description of reason for non-transmission of multidisciplinary correspondence documents in the B2 group | Hospital discharge (maximum 30 days)
Rate of patients for whom a follow-up review of proposed medication changes has been performed by the pharmacist in the B2 group | 2 months post discharge
Number of multidisciplinary correspondence documents transmitted by community pharmacist in group B2 | 2 months post hospital discharge
Rate of patients with at least one rehospitalization in each group | 3 months after hospital discharge
Mortality rate in each group | 3 months after hospital discharge
Healthcare team satisfaction in interventional groups (B1, B2) | 3 months after hospital discharge
  Custom-built 7-part questionnaire
patient satisfaction in all groups (A, B1, B2) | 3 months after hospital discharge
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Kinowski, Principal Investigator — Nîmes University Hospital
Locations (4):
- France (4):
  - Chu de Grenoble, Grenoble
  - CHU de Montpellier, Montpellier
  - Nimes University Hospital, Nîmes
  - CHU de Toulouse, Toulouse